CLINICAL TRIAL: NCT04429958
Title: The Belgian Diabetes in Pregnancy Follow-up Study
Acronym: BEDIP-FUS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); Onze Lieve Vrouw Hospital (Other); Imelda Bonheiden (Unknown)
Responsible Party: Sponsor
Other Study IDs: S64070
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Gestational Diabetes; Type2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GDM: 125 mothers with a history of GDM in pregnancy at the time of the BEDIP study and their offspring born during the BEDIP study
  Interventions: Other: GDM
- abnormal GCT group: 125 mothers with an abnormal glucose challange test (GCT of 130mg/dl or more) in pregnancy at the time of the BEDIP study and their offspring born during the BEDIP study
- normal group: 125 mothers with both a normal GCT and OGT in pregnancy at the time of the BEDIP study and their offspring born during the BEDIP study

INTERVENTIONS:
Other: GDM — different degrees of hyperglycaemia during pregnancy
  Groups: GDM

SUMMARY:
Gestational diabetes (GDM) is a form of diabetes that develops during pregnancy. GDM is associated with increased risks for pregnancy complications such as macrosomia s and preterm delivery. Women with a history of GDM have a high risk to develop a type 2 diabetes (T2DM) within the next ten years after delivery. The children are also at increased risk of developing obesity and T2DM later in life. Studies are needed to find more accurate predictors for the metabolic risk later in life. This will help to individualize the follow-up and to develop tailored prevention strategies in women and offspring with a history of GDM. In this research project we will therefore investigate how the long-term metabolic risk can more accurately be predicted in a follow-up cohort of the 'Belgian Diabetes in Pregnancy study' (BEDIP-N). We will study the relationship between maternal weight, degree of body fat and degree of hyperglycaemia in pregnancy on the long-term metabolic risk of 375 women and offspring pairs 3-7 years after the delivery across different gestational glucose tolerance groups based on the 2013 WHO criteria in pregnancy. In addition, we will study whether a promising new biomarker, glycated CD59, is a good predictor for the long-term metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who participated in the completed BEDIP-N study and received both the GCT as the OGTT during pregnancy
* Offspring born at the time of participation in the BEDIP-N study

Exclusion Criteria:

* Mothers:

  * Current pregnancy
  * Treatment that influences glycaemic status such as high dose corticoids.
  * History of bariatric surgery
  * gastro-intestinal surgery changing the absorption of glucose (Billroth II)
  * A normal study visit will not be possible (incompliance, psychiatric problems…)
  * Diagnosed with type 1 diabetes or the presence of auto-immune antibodies for type 1 diabetes

Offspring:

* Treatment that influences glycaemic status such as high dose corticoids.
* A normal study visit will not be possible (incompliance, psychiatric problems…)
* Diagnosed with type 1 diabetes or the presence of auto-immune antibodies for type 1 diabetes

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We plan to recruit 375 women-offspring pairs with the five largest centers who participated in the initial BEDIP study. Women and offspring will be recruited according to 3 different subgroups based on the antenatal result of the GCT and OGTT in the index pregnancy (a sample of 125 in each group): GDM group; normal glucose tolerance (NGT) on the OGTT with an abnormal preceding GCT (abnormal GCT NGT group); NGT on the OGTT with a normal preceding GCT (normal GCT NGT group). Abnormal GCT is defined as glucose≥130mg/dl, in line with our previous research.
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
A disorder of glucose metabolism in mothers | 3-7 years after delivery
  T2DM defined by the 75g OGTT and/or HbA1c, or prediabetes defined by the American Diabetes Association (ADA) criteria
BMI in offspring | 3-7 years after delivery
  BMI z score as a continuous variable

SECONDARY OUTCOMES:
BMI in mothers | 3-7 years after delivery
  BMI as continuous variable
metabolic syndrome in mothers | 3-7 years after delivery
  The metabolic syndrome based on the WHO criteria
Insulin sensitivity mothers Matsuda | 3-7 years after delivery
  Insulin sensitivity measured by the insulin sensitivity index of Matsuda
Insulin sensitivity mothers HOMA | 3-7 years after delivery
  Insulin sensitivity measured by the reciprocal of the homeostasis model assessment of insulin resistance (1/HOMA-IR)
Beta-cell function mothers HOMA-B | 3-7 years after delivery
  Beta-cell function by the HOMA-B index and the insulinogenic index divided by HOMA-IR
Beta-cell function mothers ISSI-2 | 3-7 years after delivery
  Beta-cell function measured by the insulin-secretion sensitivity-2 index
Beta-cell function mothers Stumvoll | 3-7 years after delivery
  Beta-cell function measured by the Stumvoll index
Adiposity mothers BIA | 3-7 years after delivery
  Adiposity (as a continuous variable) measured by the bioelectrical impedance analysis
Adiposity mothers skin folds | 3-7 years after delivery
  Adiposity (as a continuous variable) measured by skin folds
overweight offspring | 3-7 years after delivery
  overweight defined by BMI z score according to the WHO guidelines
obesity offspring | 3-7 years after delivery
  obesity defined by BMI z score according to the WHO guidelines
A disorder of glucose metabolism in offspring | 3-7 years after delivery
  T2DM and prediabetes based on the fasting plasma glucoseand/or HbA1c defined by the ADA criteria
metabolic syndrome in offsping | 3-7 years after delivery
  metabolic syndrome based on the WHO criteria
insulin sensitivity offspring | 3-7 years after delivery
  insulin sensitivity measured by HOMA-IR
Beta-cell function offsping | 3-7 years after delivery
  Beta-cell function by the HOMA-B index
Adiposity offsping BIA | 3-7 years after delivery
  Adiposity (as a continuous variable) measured by the bioelectrical impedance analysis
Adiposity offsping skin folds | 3-7 years after delivery
  Adiposity (as a continuous variable) measured by skin folds

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Benhalima, Principal Investigator — UZ Leuven
Locations (5):
- Belgium (5):
  - OLV-Alast, Aalst
  - UZA, Antwerp
  - OLV-Asse, Asse
  - Imelda Bonheiden, Bonheiden
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No